CLINICAL TRIAL: NCT06693154
Title: A Comparative Study of Serum and Fecal Calprotectin Levels in Necrotizing Enterocolitis
Brief Title: Calprotectin Levels in Necrotizing Enterocolitis
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Sara EROL, Assoc Prof, MD, Ankara Yildirim Beyazıt University
Other Study IDs: 26379996/26, 03-2022
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Necrotising Enterocolitis Neonatal
Keywords: calprotectin; necrotising enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 59 Days
Biospecimen Retention: Samples Without DNA — Fecal and blood samples were collected from each eligible patient and were immediately stored at -20°C until batch analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Premature infants diagnosed with stage 2 and stage 3 NEC and a matched control group.

SUMMARY:
Necrotizing enterocolitis (NEC) is a serious condition that can affect premature babies, leading to complications like intestinal damage and infection. In our study, we measured specific markers (called calprotectin) in blood and stool to understand how severe NEC is and predict outcomes. We found that these markers were higher in babies with more severe NEC (stage 3), especially in those who needed surgery or sadly did not survive. This information can help doctors detect NEC earlier, understand its severity, and make better decisions for treating affected babies.

ELIGIBILITY:
Inclusion Criteria:

before 32 weeks of gestation with a birth weight of ≤1500 grams

Exclusion Criteria:

Infants whose families did not provide consent and those with congenital anomalies were excluded.

Ages: 3 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns admitted to the neonatal intensive care unit (NICU) over a 2-year period, born at or before 32 weeks of gestation with a birth weight of ≤1500 grams, were included in this study.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
The predictive value of serum and fecal calprotectin levels in necrotising enterocolitis (NEC) | 2 years
  The predictive value of serum and fecal calprotectin levels in assessing NEC severity (stage 2 and stage 3), intestinal perforation, the need for surgery, and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Kurt, Study Director — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: The IPD and supporting information will be available starting 6 months after the publication of the study results and will remain one year.
Access Criteria: Access to IPD and supporting information will be available to qualified researchers affiliated with academic or medical institutions. They will be able to access study protocol through a formal data-sharing agreement. Requests must be submitted via email to [sarasurmeli@gmail.com]

REFERENCES:
- [Derived] Erol S, Tayman C, Korkut S, Cakir U, Kurt A, Koyuncu I. A comparative study of serum and fecal calprotectin levels in necrotizing enterocolitis. J Pediatr (Rio J). 2025 Sep-Oct;101(5):101428. doi: 10.1016/j.jped.2025.101428. Epub 2025 Aug 21. PMID 40784368